CLINICAL TRIAL: NCT07345299
Title: Development and Measurement of the Effects of a Digital Education Solution for Patients Undergoing Total Hip or Knee Arthroplasty
Acronym: CHUVeduc@home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole de Santé Vaud (Other)
Responsible Party: Principal Investigator, Claude Pichonnaz, Associate Professor UAS, Ph.D, Haute Ecole de Santé Vaud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUVeduc@home
Record Dates: First submitted 2025-08-29; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty Replacement, Knee; Arthroplasty, Replacement, Hip
Keywords: knee; hip; replacement; arthroplasty; patient education; digital solution; preoperative care; perioperative care; interdisciplinary intervention; physiotherapy; nursing; health literacy; digital literacy

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: access to CHUVeduc@home before surgery (Experimental): Intervention Group - Pathway with CHUVeduc@home This group follows the standard preoperative pathway, complemented by personalized digital preparation through the CHUVeduc@home application, available 2 to 6 weeks before surgery.
  Interventions: Behavioral: Digital Preoperative Education with CHUVeduc@home
- Control Group - Standard Care Pathway (Active Comparator): Control Group - Standard Care Pathway This group follows the standard clinical care pathway established at CHUV for patients undergoing total hip or knee arthroplasty.
  The main steps include:
  * Consultation with the surgeon
  * Group information session
  * Preoperative consultation
  * Hospital stay for surgery
  * Discharge and return home
  * Telemonitoring with CHUV@home after surgery
  * Postoperative follow-up visit at 6 weeks
  Participants in this group also use the CHUV@home application to complete study-specific questionnaires; however, they do not receive any additional educational content prior to surgery.
  Interventions: Behavioral: Standard Care Pathway

INTERVENTIONS:
Behavioral: Digital Preoperative Education with CHUVeduc@home — The intervention consists of a personalized digital education program delivered through the CHUVeduc@home mobile application, integrated within the existing CHUV@home platform. The application is available to patients 2 to 6 weeks prior to surgery and provides:
  * Educational modules covering postoperative recovery, pain management, rehabilitation, and discharge planning.
  * Quizzes and knowledge tests to reinforce patient understanding.
  * Practical advice sheets for concrete preparation.
  * Individualized pacing and guidance tailored to patient needs.
  * Notifications prompting completion of study questionnaires.
  The goal of the intervention is to improve patient health literacy, reduce preoperative anxiety, increase confidence, and facilitate recovery and return home after total hip or knee arthroplasty.
  Arms: Intervention Group: access to CHUVeduc@home before surgery
Behavioral: Standard Care Pathway — The main steps include:
  * Consultation with the surgeon
  * Group information session
  * Preoperative consultation
  * Hospital stay for surgery
  * Discharge and return home
  * Telemonitoring with CHUV@home after surgery
  * Postoperative follow-up visit at 6 weeks
  Participants in this group also use the CHUV@home application to complete study-specific questionnaires; however, they do not receive any additional educational content prior to surgery.
  Arms: Control Group - Standard Care Pathway

SUMMARY:
This study aims to evaluate the effectiveness of a digital patient education solution, CHUVeduc@home, in improving preoperative preparation for patients undergoing total hip or knee arthroplasty. In Switzerland, many patients receive joint replacements each year to relieve osteoarthritis-related pain. With shorter hospital stays, adequate preparation before surgery has become increasingly important.

A total of 160 patients will be randomized into two groups:

Intervention group: access to CHUVeduc@home before surgery. Control group: standard preoperative preparation (group information session and consultation).

All participants will complete questionnaires through the application. No additional visits are required. The intervention lasts approximately 12 weeks.

The primary goal is to determine whether digital education increases patient knowledge, confidence, and satisfaction, and facilitates recovery and return home after surgery. Participation is voluntary and can be withdrawn at any time.

DETAILED DESCRIPTION:
Study Purpose:

The purpose of this study is to improve preparation for hip or knee surgery. Each year in Switzerland, a large number of individuals receive a hip or knee prosthesis to relieve pain caused by osteoarthritis. Through enhanced perioperative care programs such as the one implemented at CHUV, the length of hospital stay has decreased, making preoperative preparation increasingly important.

Current Practice:

Current practice includes participation in a group information session and a preoperative consultation. However, retaining all provided information can be challenging. To support more effective preparation, the investigators will evaluate a digital application called CHUVeduc@home, integrated within CHUV@home, which is already used during postoperative recovery.

Features of the Application:

The application provides the possibility to:

Review information at an individualized pace. Improve understanding of the surgical and recovery processes. Access quizzes and practical information sheets for training purposes.

Submit questions directly to the Telemonitoring Center team.

Study Design:

The study plans to include 160 participants. Participants will be randomly assigned to one of two groups:

A group using the application before surgery. A group following the usual preoperative preparation process.

All participants will use the application to complete study questionnaires. No additional appointments are required. The study duration is approximately 12 weeks. Participation is voluntary and can be discontinued at any time.

Expected Benefits:

The investigators anticipate that this digital approach to preoperative preparation may help participants feel more confident, better informed, and better supported during their return home after surgery.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients admitted to the CHUV musculoskeletal department during the study period
* primary total hip replacement or primary total knee replacement
* a Risk Assessment and Prediction Tool (RAPT) score >6

Exclusion Criteria:

* a RAPT score <6,
* knee/hip arthroplasty revision surgery
* inability to give informed consent or answer questionnaires knowledgeably due to language or cognitive impairment as reported in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patient calls to the remote care center (CTS) | During the intervention period (from inclusion until surgery, up to 6 weeks)
  The primary outcome is the total number of calls initiated by patients to the remote care support center (CTS) during the intervention period. This measure will assess the impact of the digital education tool on patient autonomy and the need for additional support. A lower number of calls is expected to reflect improved patient preparation and self-management.
Reason for contacts, the severity of alerts | During the intervention period (from inclusion until surgery, up to 6 weeks)
  This secondary objective aims to analyze the specific reasons for patient contacts, assess the severity of alerts generated, and evaluate the potential financial benefits associated with a decrease in the number of contacts, thereby providing a comprehensive understanding of the impact of the telemonitoring intervention.

SECONDARY OUTCOMES:
Patient-reported health status and quality of life (EQ-5D-5L) | At preadmission (3 days before surgery), and 6 weeks postoperatively
  Generic health-related quality-of-life measure including five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and a visual analogue scale (VAS).
  Range:
  Index score: typically ranges from <0 (health states worse than death) to 1 (perfect health).
  VAS: 0 to 100, where 100 indicates the best imaginable health.
  Direction: Higher scores reflect better health status.
Patient satisfaction (ANQ questionnaire) | 1 week after hospital discharge
  Patient satisfaction with hospital care will be evaluated using the Association Nationale pour la Qualité (ANQ) patient satisfaction questionnaire.
  The ANQ questionnaire includes multiple items each rated on a Likert scale from 1 to 5, where higher scores indicate greater satisfaction. Depending on the domain structure used locally, total scores typically range from 1 (lowest satisfaction) to 5 (highest satisfaction) per item; domain or global scores are expressed as mean values, with higher values reflecting better satisfaction with care.
Patient engagement (Patient Activation Measure [PAM-13] | At baseline during the intervention period , at preadmission (3 days before surgery) and 6 weeks postoperatively
  Patient engagement in disease management and surgical preparation will be assessed using the Patient Activation Measure-13 (PAM-13).
  The PAM-13 contains 13 items, each scored from 1 (strongly disagree) to 4 (strongly agree).
  Raw scores are converted to a standardized activation score ranging from 0 to 100.
  Higher scores indicate greater patient activation, confidence, and involvement in their own health management.
  Scores classify patients into four activation levels, with Level 1 = lowest activation and Level 4 = highest activation.
Physical activity (International Physical Activity Questionnaire [IPAQ]) | At baseline during the intervention period and 6 weeks postoperatively
  Physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ - Short Form).
  The IPAQ evaluates physical activity performed in the last 7 days across four domains: walking, moderate-intensity activity, vigorous-intensity activity, and sedentary time.
  Scores are expressed as Metabolic Equivalent of Task (MET)-minutes per week. Total physical activity score typically ranges from 0 MET-min/week (no reported activity) to > 3,000 MET-min/week (very high activity levels).
  Higher MET-min/week scores indicate higher levels of physical activity.
  Participants will also be classified into the IPAQ categories:
  Low physical activity, Moderate physical activity, High physical activity, based on standard IPAQ scoring guidelines.
Fear and anxiety related to surgery (Survey of Surgical Fear [SSF]) | At baseline during the intervention period and at preadmission (3 days before surgery)
  Fear and anxiety associated with the upcoming surgery will be measured using the Survey of Surgical Fear (SSF).
  The SSF includes 8 items, each rated from 0 (not at all fearful) to 10 (extremely fearful).
  Total score range: 0 to 80.
  The questionnaire provides two subscale scores:
  * Short-term surgical fear (items 1-4), range 0-40
  * Long-term surgical fear (items 5-8), range 0-40
  Higher scores indicate higher levels of fear and anxiety related to surgery.
Pain (Numeric Rating Scale for pain) | At hospital discharge (Day 3-5) and at 6 weeks postoperatively
  Patients will report pain intensity using the Numeric Rating Scale (EVA), during routine follow-up visits.
Patients' expectations regarding surgery outcomes (Hospital for Special Surgery Knee/Hip Expectations Survey [HSS Knee or Hip]) | At baseline (prior to surgery) during the intervention period
  Patient expectations concerning pain relief, mobility, essential daily activities, psychological benefits, and non-essential activities (e.g., sport/leisure) will be measured using the Hospital for Special Surgery (HSS) Knee or Hip Expectations Survey, depending on the type of surgery.
Qualitative analysis of patient messages to the remote care team (CTS) | During the intervention period (from inclusion until surgery, up to 12 weeks)
  A qualitative review of the messages sent by patients to the remote care support team (CTS) will be performed to identify difficulties encountered during the intervention and the solutions provided.
Patient-reported Oxford Knee Score [OKS] or Oxford Hip Score [OHS]) | At preadmission (3 days before surgery) and 6 weeks postoperatively
  Joint-specific questionnaire assessing knee or hip pain and functional ability after knee or hip surgery.
  Range: 0 to 48, based on 12 items (0-4 per item).
  Direction: Higher scores indicate better knee or hip function and less pain.
Patient satisfaction with mobile application (uMARS scale) | At preadmission (3 days before surgery)
  Satisfaction with the mobile application will be assessed using the User Version of the Mobile Application Rating Scale (uMARS).
  The uMARS consists of 20 items rated from 1 to 5, grouped into four objective quality subscales (engagement, functionality, aesthetics, information) and one subjective quality subscale. Subscale and total scores range from 1 (poor quality) to 5 (excellent quality). Higher uMARS scores reflect greater perceived app quality and satisfaction.
Health literacy, French eHealth Literacy Scale [F-eHEALS]) | At baseline during the intervention period and 6 weeks postoperatively
  Health literacy will be evaluated using the French version of the eHealth Literacy Scale (F-eHEALS).
  The F-eHEALS contains 8 items, each rated from 1 (strongly disagree) to 5 (strongly agree).
  Total score range: 8 to 40. Higher scores indicate better perceived eHealth literacy, including ability to find, appraise, and use online health information.
Postoperative complications (clinical assessment) | At hospital discharge (Day 3-5) and at 6 weeks postoperatively
  Postoperative complications will be recorded by clinical staff according to routine medical documentation.
  Outcomes include the presence or absence of complications and the type of complication (e.g., infection, thromboembolic event, wound complication, cardiovascular or respiratory event).
  This is a categorical clinical outcome (no scoring scale).
Length of stay (days of hospitalization) | At hospital discharge
  Length of hospital stay, expressed in days, with higher values indicating longer hospitalization.
Hospital readmission (yes/no) | At 6 weeks postoperatively
  Hospital readmissions within the follow-up period will be recorded by clinical staff.
  Reported as yes/no, with reason for readmission documented when applicable. This is a binary clinical outcome (no scoring scale).
Stratified analysis of intervention effectiveness by patient characteristics | At the end of the intervention period (up to 12 weeks after inclusion)
  A stratified analysis will be conducted to evaluate whether the impact of the digital education intervention varies across patient subgroups (e.g., age, education level, comorbidity profile). This will help identify clusters of patients who benefit most from digital education.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichonnaz, Ph.D, Principal Investigator — Haute Ecole de Santé Vaud
Locations (1):
- University Hospital of Lausanne CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agri F, Hahnloser D, Demartines N, Hubner M. Gains and limitations of a connected tracking solution in the perioperative follow-up of colorectal surgery patients. Colorectal Dis. 2020 Aug;22(8):959-966. doi: 10.1111/codi.14998. Epub 2020 Feb 27. PMID 32012423
- [Background] Roulin D, Blanc C, Demartines N, Hubner M. [Enhanced Recovery After Surgery--optimal management of the surgical patient]. Rev Med Suisse. 2014 Jun 18;10(435):1343-7. French. PMID 25051597
- [Background] Ljungqvist O, Hubner M. Enhanced recovery after surgery-ERAS-principles, practice and feasibility in the elderly. Aging Clin Exp Res. 2018 Mar;30(3):249-252. doi: 10.1007/s40520-018-0905-1. Epub 2018 Feb 16. PMID 29453605
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- See also: SIRIS Swiss National Joint Registry, Hip and Knee 2023 — https://www.siris-implant.ch/fr/Downloads&category=16
- See also: CHUV@home : pour faciliter le suivi des patients à domicile 2020 — https://www.chuv.ch/fr/pratique/informations-pratiques/offre/web_ofr_75/application-chuvhome
- See also: Health Literacy Survey Schweiz 2019-2021 — https://www.sages.ch/wp-content/uploads/2021/09/HLS19-21-CH_Schlussbericht_Careum-Gesundheitskompetenz_Health-Literacy-Survey_20210914-1.pdf
- See also: Compétences en matière de cybersanté: Office fédéral de la santé publique; 2019 — https://www.e-health-suisse.ch/fr/coordination/informations/formation-et-habilitation